CLINICAL TRIAL: NCT00149877
Title: Efficacy, Safety and Tolerability of Tegaserod in Patients With Chronic Constipation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CHTF919EHK01
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2008-02-01 (Estimated); Status verified 2008-01

CONDITIONS: Chronic Constipation
Keywords: Chronic constipation, tegaserod
MeSH Terms: interventions — tegaserod

INTERVENTIONS:
Drug: Tegaserod

SUMMARY:
Tegaserod (HTF919) is an aminoguanidine indole compound and a member of a new class of subgroup-selective 5-hydroxytryptamine (5-HT) agonists. The aim of this study is to investigate the efficacy, safety and tolerability of tegaserod on bowel habits in patients with CC.

ELIGIBILITY:
Inclusion Criteria:

* Male and females of at least 18 years of age
* A 12-month history of constipation (defined as < three spontaneous bowel movements per week and ≥1 of the following symptoms >25% of the time: hard stools, sensation of incomplete evacuation and straining)

Exclusion Criteria:

* Patients with cancer, inflammatory bowel disease or other structural bowel disease
* Patients who participated in a prior tegaserod study
* Evidence of cathartic colon or laxative abuse, pelvic floor dysfunction or neurological disorders

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-04; Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Number of complete spontaneous bowel movement (csbm) during the first 4 weeks of treatment.

SECONDARY OUTCOMES:
Number of csbm during 8 weeks of treatment.
Daily assessment of bowel habits:frequency, form, straining, feeling of complete evacuation.
Daily patients' assessment: bowel habits, constipation, distention/bloating, abdominal discomfort pain.
Laxative use.
Safety and tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Basel
Locations (1):
- Novartis, Basel, Switzerland